CLINICAL TRIAL: NCT00726414
Title: A Relative Bioavailability Study of Quinine Sulfate Capsules 324mg Under Fasting and Fed Conditions
Brief Title: A Relative Bioavailability Study of Quinine Sulfate Capsules 324mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Matthew Davis, M.D., Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R05-1613
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2010-02-03 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quinine Sulfate Capsules 2 x 324 mg Capsules - Fasting (Experimental): A single dose of Quinine Sulfate (2 x 324 mg capsules) administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Quinine Sulfate 2 x 324 mg Capsules
- Quinine Sulfate Capsules 2 x 324 mg Capsules - Fed (Experimental): A single dose of Quinine Sulfate (2 x 324 mg capsules) administered 30 minutes after a standardized, high fat breakfast.
  Interventions: Drug: Quinine Sulfate 2 x 324 mg Capsules

INTERVENTIONS:
Drug: Quinine Sulfate 2 x 324 mg Capsules — Quinine Sulfate (2 x 324 mg capsules) administered after an overnight fast of at least 10 hours.
  Arms: Quinine Sulfate Capsules 2 x 324 mg Capsules - Fasting
Drug: Quinine Sulfate 2 x 324 mg Capsules — Quinine Sulfate (2 x 324 mg capsules) administered 30 minutes after a standardized, high fat breakfast.
  Arms: Quinine Sulfate Capsules 2 x 324 mg Capsules - Fed

SUMMARY:
The purpose of this study is to evaluate and compare the relative bioavailability of Quinine Sulfate capsules following a single, oral dose in healthy volunteers under fasting and fed conditions.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the relative bioavailability of Quinine Sulfate capsules following a single, oral dose in healthy volunteers under fasting and fed conditions.

Twenty-two healthy, non-smoking, non-obese, male and female volunteers between the ages of 18 and 45 years of age will be randomly assigned in a crossover fashion to receive each of two Quinine Sulfate dosing regimens in sequence with a 7 day washout period between dosing periods. On the morning of Day 1, subjects will receive either a single oral dose of Quinine Sulfate (2 x 324 mg capsules) following an overnight fast of at least 10 hours, or a single oral dose of Quinine Sulfate (2 x 324 mg capsules) 30 minutes after a standardized, high-fat breakfast. After a 7 day washout period, on the morning of Day 8, subjects will receive the alternate regimen. Blood samples will be drawn from all participants before dosing and for 48 hours post-dose to adequately define the pharmacokinetics of Quinine Sulfate. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drug and/or procedures. Blood pressure and heart rate will be measured prior to dosing and at 1, 2, 4 and 12 hours after each dose and at study exit. A 12 lead electrocardiogram (EKG) will be recorded at study check-in and at 2, 4, 6, 12 and 24 hours after dose administration. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers selected for this study will be healthy men and women 18 to 45 years of age at the time of dosing. Weight range will not exceed ±20% for height and body frame
* Screening Procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and human immunodeficiency virus (HIV) antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures
* Screening will include general observations, physical examination, demographics, medical history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems
* Screening Procedures:
* Hematology: hematocrit, hemoglobin, white blood cell (WBC) count with differential, red blood cell (RBC) count, platelet count
* Clinical chemistry: serum creatinine, blood urea nitrogen (BUN), glucose, AST(SGOT - Serum glutamic-oxaloacetic transaminase), ALT(SGPT - Serum glutamic-pyruvic transaminase), albumin, total bilirubin, total protein, and alkaline phosphatase
* HIV antibody, hepatitis B surface antigen, hepatitis C antibody screens
* Urinalysis: by dipstick; full microscopic examination if dipstick positive; and
* Urine drug screen: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine
* Serum pregnancy screen (female volunteers only)
* If female and:
* of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condom with spermicide, diaphragm with spermicide, intrauterine device (IUD), or abstinence; or
* is postmenopausal for at least 1 year; or
* is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse
* Volunteers with a presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by clinical investigators)
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant
* Volunteers demonstrating a reactive screen for hepatitis B surface antigen, hepatitis C antibody or HIV antibody
* Volunteers demonstrating a positive drug abuse screen when screened
* Female volunteers demonstrating a positive pregnancy screen
* Female volunteers who are currently breastfeeding
* Volunteers with a history of allergic response(s) to quinine or related drugs
* Volunteers with a history of clinically significant allergies including drug allergies
* Volunteers with a clinically significant illness during the last 4 weeks prior to Period I dosing (as determined by the clinical investigators)
* Volunteers who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study
* Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study
* Volunteers who report receiving any investigational drug within 28 days prior to Period I dosing
* Volunteers who report taking any systemic prescription medication in the 14 days prior to Period I dosing
* Volunteers who currently use tobacco products
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing
* Male volunteers with a corrected QT interval (QTc)> 430 milliseconds (msec)on the screening electrocardiogram (ECG) or with clinically significant findings
* Female volunteers with a QTC> 450 msec on the screening ECG or with clinically significant findings

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2005-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Quinine Sulfate Under Fasted Then Fed Conditions: On the morning of Day 1 subjects received one dose of Quinine Sulfate (2 x 324 mg capsules) after an overnight fast of at least 10 hours, followed by a 7 day washout period. On the morning of Day 8 subjects received one dose of Quinine Sulfate (2 x 324 mg capsules) 30 minutes following a standardized, high fat breakfast.
- Quinine Sulfate Under Fed Then Fasted Conditions: On the morning of Day 1 subjects received one dose of Quinine Sulfate (2 x 324 mg capsules) 30 minutes following a standardized, high fat breakfast, followed by a 7 day washout period. On the morning of Day 8 subjects received one dose of Quinine Sulfate (2 x 324 mg capsules) following an overnight fast of at least 10 hours.
Period: First Intervention
Arm/Group | Quinine Sulfate Under Fasted Then Fed Conditions | Quinine Sulfate Under Fed Then Fasted Conditions
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Quinine Sulfate Under Fasted Then Fed Conditions | Quinine Sulfate Under Fed Then Fasted Conditions
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Quinine Sulfate Under Fasted Then Fed Conditions | Quinine Sulfate Under Fed Then Fasted Conditions
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Quinine Sulfate Under Fed and Fasted Conditions: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one dose of Quinine Sulfate (2 x 324 mg capsules) following an overnight fast or 30 minutes following a standardized, high fat breakfast.
Arm/Group | Quinine Sulfate Under Fed and Fasted Conditions
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 20.6 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) for Quinine Sulfate
Description: The maximum or peak concentration that Quinine Sulfate reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hours after drug administration.
Population: Data from all 22 subjects enrolled in this study were used in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Quinine Sulfate Under Fasted Conditions: Each subject received two capsules of Quinine Sulfate 324 mg after an overnight fast of at least 10 hours.
- Quinine Sulfate Under Fed Conditions: Each subject received two capsules of Quinine Sulfate 324 mg 30 minutes following a standardized, high fat breakfast.
Arm/Group | Quinine Sulfate Under Fasted Conditions | Quinine Sulfate Under Fed Conditions
Number analyzed (Participants) | 22 | 22
ng/mL | 3,293.84 (750.85) | 3,424.30 (859.91)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)] for Quinine Sulfate
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: Data from all 22 subjects enrolled in this study were used in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Quinine Sulfate Under Fasted Conditions | Quinine Sulfate Under Fed Conditions
Number analyzed (Participants) | 22 | 22
ng-hr/mL | 49,484.64 (15,831.86) | 51,228.07 (16,690.68)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)] for Quinine Sulfate
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: Data from all 22 subjects enrolled in this study were used in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Quinine Sulfate Under Fasted Conditions | Quinine Sulfate Under Fed Conditions
Number analyzed (Participants) | 22 | 22
ng-hr/mL | 52,643.14 (18,056.00) | 54,409.12 (18,706.05)

ADVERSE EVENTS:
Arm/Group | Quinine Sulfate Under Fasted Conditions | Quinine Sulfate Under Fed Conditions
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 4/22 | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinine Sulfate Under Fasted Conditions (N=22) | Quinine Sulfate Under Fed Conditions (N=22)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dysmenorrhea (Endocrine disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days